CLINICAL TRIAL: NCT06807125
Title: Intraoral Wear Measurement of Opposing Enamel to Indirect Milled Resin Matrix Ceramic Versus Direct Bulk Fill Resin Composite in Posterior Teeth After Using 2 Years: Randomized Clinical Trial
Brief Title: Wear Measurement of Opposing Enamel to Milled Resin Matrix Ceramic Versus Bulk Fill Resin Composite After 2 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Esraa Esmeail Hussien, Lecturer, Misr University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-0063
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Dental Wear
Keywords: Wear measurements, resin matrix ceramic, Bulk fill composite, Digital scanner.
MeSH Terms: conditions — Tooth Wear

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding empowers the research to minimize threats to internal validity and strengthen the external validity. Our clinical trial was double blinding, the participant and the outcomes assessor were blinded while, the investigator cant be blinded as he worked with two different materials and techniques
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resin matrix ceramic block (Experimental): BRILLIANT Crios is the ideal choice for single-tooth restorations, both in the anterior and the posterior region. It is composed of dental glass (barium glass ˂ 1.0 μm), amorphous silica (Sio2 ˂ 20 nm), resin matrix (cross-linked methacrylates) and pigments (inorganic pigments such as ferrous oxide or titanium dioxide).
  Interventions: Procedure: Resin matrix ceramic block
- Direct Restoration (Active Comparator): 3M™ Filtek™ One Bulk Fill Restorative is a visible light activated, restorative composite optimized to create fast and easy restorations. The material can be placed and cured up to 5 mm deep, enabled by a stress relieving resin system and optimized optical properties. It is composed of fillers which are a combination of a non-agglomerated/non-aggregated 20 nm silica filler.
  4 to 11 nm zirconia filler, zirconia/silica cluster filler and ytterbium trifluoride filler consisting of 100nm particles. The inorganic filler loading is about 76.5% by weight (58.5% by volume). It contains AFM (dynamic stress-relieving monomer), AUDMA, UDMA and 1, 12-dodecane-DMA. 3M™ Filtek™ Bulk Fill Posterior Restorative is applied to the tooth following use of a methacrylate-based dental adhesive
  Interventions: Procedure: Resin matrix ceramic block

INTERVENTIONS:
Procedure: Resin matrix ceramic block — Milled resin composite block for fabrication of permanent, indirect restorations using a CAD/CAM grinding process. shock absorbing affect due to the dentin- like modulus of elasticity makes BRILLIANT Crios will suited or indirect restoration.
  Other Names: CAD/CAM Reinforced composite overlay

SUMMARY:
This clinical trial conducted to measure the amount of wear of opposing enamel to indirect milled resin matrix ceramic versus direct bulk fill resin composite intraorally using Digital Scanner after two years of using

DETAILED DESCRIPTION:
Indirect milled resin matrix ceramic overlay versus direct bulk fill resin composite overlay was utilized in a clinical trial to compare the amount of enamel wear on endodontically treated molars using a Panda P2 digital scanner and Geomagic Control X 3D software. After one and two years, measurements of enamel wear were taken.

ELIGIBILITY:
Inclusion Criteria:

* ● Patients with non vital badly decayed posterior teeth.

  * 18 -55years.
  * Males or Females.
  * Good oral hygiene.
  * Co-operative patients approving to participate in the study

Exclusion Criteria:

* High caries index.

  * Severe medical complications.
  * Pregnancy.
  * Allergic history concerning methacrylates Disabilities.
  * Heavy smoking.
  * Xerostomia.
  * Lack of compliance.
  * Evidence of parafunctional habits.
  * Temporomandibular joint disorders.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Amount of Enamel Wear | two years follow up
  amount of enamel wear measured through superimposition of STL files exported from intraoral scanner then using geomagic Control X 3D

CONTACTS AND LOCATIONS:
Overall Officials: Esraa EE Hussien, PhD, Principal Investigator — Misr University for Science and Technology
Locations (1):
- Misr University for Science and Technology, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No